CLINICAL TRIAL: NCT07338435
Title: "Comparison of Preservation Residual Renal Function and Oxidative Damage Between Incremental and Standard Peritoneal Dialysis in Incident Patients at Two Centers of Mexico.
Brief Title: "Residual Kidney Function and Oxidative Stress in Incremental vs Standard Peritoneal Dialysis (2 Mexican Centers)"
Acronym: INSPiRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Veronica Valdivia Cerda, Clinical prophesor, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R-2024-1009-44
Record Dates: First submitted 2025-11-25; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Diabetic Kidney Disease; Peritoneal Dialysis (PD); Hypertension; Hypertension With Renal Dysfunction
Keywords: inflammation.; chronic kidney disease.; oxidative stress; malondialdehyde; residual kidney function; incremental peritoneal dialysis; peritoneal dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies; Hypertension; Inflammation

STUDY DESIGN:
Intervention Model Description: The researchers will assign the participants by lottery using a table of numbers to each of the incremental or standard dialysis treatments, forming groups A and B.
  To form the treatment groups, the options will be A: Incremental peritoneal dialysis (IPD) and B: Standard peritoneal dialysis (standard PD or CAPD). A probabilistic number will be determined using block randomization, so the group will be divided into 10 blocks of 4 patients each, assigning 2 to group A and 2 to group B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental peritoneal dialysis (IPD) (Experimental): uses reduced dialysis doses less exchanges, generally 3 or less
  Interventions: Procedure: Incremental Peritonal Dialysis
- Standard peritoneal dialysis (SPD) (Active Comparator): standard peritoneal dialysis (SPD)-which typically involves four daily exchanges of 4-5 hours each one with night exchange, known too like full-dose dialysis
  Interventions: Procedure: Standard Peritoneal Dialysis

INTERVENTIONS:
Procedure: Standard Peritoneal Dialysis — 4 exchanges with nocturnal dwell.
  Other Names: DPCA
  Arms: Standard peritoneal dialysis (SPD)
Procedure: Incremental Peritonal Dialysis — lower dialysis doses based on RKF, generally 3 exchanges or less.
  Other Names: IPD
  Arms: Incremental peritoneal dialysis (IPD)

SUMMARY:
Title:

Comparison of Oxidative Stress and Preservation of Residual Kidney Function Between Incremental and Standard Peritoneal Dialysis in Incident Patients at the Regional General Hospital No. 58 and HGZ/UMF 21 of the Mexican Institute of Social Security (IMSS) in León, Guanajuato

BACKGROUND:

Peritoneal dialysis (PD) employs hypertonic dextrose-based solutions to remove toxins and excess fluids. This exposure promotes mitochondrial overproduction of reactive oxygen species (ROS), triggers inflammation, and may accelerate the decline of residual kidney function (RKF), leading to complications such as peritonitis, peritoneal fibrosis, and technique failure. Although more biocompatible solutions are available, their high cost and limited accessibility restrict their use in our setting.

Incremental peritoneal dialysis (IPD), in contrast to standard peritoneal dialysis (SPD)-which typically involves four daily exchanges with full-dose dialysis-uses reduced dialysis doses tailored to RKF, thereby decreasing glucose exposure.

The primary aim of this study was to compare the effects of IPD versus SPD on oxidative stress, inflammation, and the preservation of residual kidney function in incident peritoneal dialysis patients at the Regional General Hospital No. 58 in León, Guanajuato.

MATERIALS AND METHODS:

A prospective, longitudinal, single-center, open-label, randomized clinical trial will be conducted. Incident peritoneal dialysis patients at the Regional General Hospital No. 58 and Gneral Hospital of Zone Numbre 21 of the Mexican Institute of Social Security (IMSS) who meet the inclusion criteria and provide informed consent will be randomly assigned to either the standard or incremental peritoneal dialysis group.

Acute-phase reactants will be measured at baseline and at 3, 6, 9, and 12 months. Oxidative stress will be assessed via baseline and end-of-study malondialdehyde levels. Dialysis and urine Kt/V will be evaluated betwen 6 weeks and 3 moths and 6, 9, and 12 months. Appropriate statistical analyses will be performed thereafter.

DETAILED DESCRIPTION:
Eligible incident peritoneal dialysis (PD) patients from two IMSS hospitals in León, Guanajuato (HGR No. 58 and HGZ-MF No. 21) will be enrolled after confirmation of adequate Tenckhoff catheter placement and written informed consent. Baseline demographic and clinical data will be collected from medical records and physical examination, including age, sex, marital status, educational level, anthropometric parameters (weight, height, body mass index), and volume status assessed by physical examination using the Godet edema scale.

Laboratory evaluations will be performed in blood and urine. Fasting venous blood samples will be obtained for complete blood count, serum chemistry, electrolytes, lipid profile, inflammatory markers (albumin, ferritin, C-reactive protein, D-dimer), and viral serology (HBV, HCV, HIV). Oxidative stress will be assessed in serum by measuring thiobarbituric acid-reactive substances (TBARS) as an index of malondialdehyde concentration using a standardized spectrophotometric method.

Residual renal function will be assessed at baseline and during follow-up (45 days, and 3, 6, 9, and 12 months) by estimated glomerular filtration rate (CKD-EPI equation), 24-hour urine volume, and 24-hour creatinine clearance. Solute clearance adequacy (renal and peritoneal Kt/V) will be measured at 1.5-3 months, 6 months, and 12 months. Peritoneal membrane transport characteristics will be evaluated at month 3 using the Peritoneal Equilibration Test (PET).

Participants will be randomized in a 1:1 ratio to Incremental Peritoneal Dialysis or Standard Peritoneal Dialysis using block randomization (blocks of four). Glucose exposure will be quantified based on dialysate glucose concentration and number of exchanges, expressed as bags per year. Catheter-related complications and infection-free catheter survival will be monitored throughout the 12-month follow-up. After completion of follow-up, patients will continue PD according to their treating nephrologist's prescription.

ELIGIBILITY:
Inclusion Criteria:

CKD adults starting on PD FKR ≥2 mL/min Urine Volumen ≥500 mL/24 hrs Type 2 Diabetes, Hypertension and unknown cause of CKD

Exclusion Criteria:

Self-reported smoking or active use of illicit drugs. Patients with liver disease. Patients with glomerulonephritis. Patients with a history of previous renal replacement therapy (hemodialysis or kidney transplant).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress Serum malondialdehyde (MDA) levels | Baseline and 12 months
  Oxidative stress will be assessed by serum malondialdehyde (MDA) concentration measured as thiobarbituric acid-reactive substances (TBARS) using spectrophotometry at 532 nm. Results will be expressed in nmol/mL.
Residual kidney function | Baseline, 45 days, 3 months, 6 months, 9 months, and 12 months
  Residual kidney function will be evaluated by estimated glomerular filtration rate (eGFR) calculated using the CKD-EPI equation (mL/min/1.73 m²), 24-hour, 24-hour urine volume (liters), and 24-hour creatinine clearance (mL/min).

SECONDARY OUTCOMES:
Systemic inflammation: Inflammatory biomarkers | at 3, 6,9, and 12 moths
  Systemic inflammation will be assessed by serum levels of C-reactive protein (CRP, mg/L), ferritin (ng/mL), albumin (g/dL), and D-dimer (ng/mL), measured using standardized laboratory methods.
Catheter-related outcomes | Up to 12 months
  Catheter outcomes will be assessed by time to first catheter-related complication or infection, expressed as complication-free catheter survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Database and Informed consent
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting documents will be available starting 6 months after publication of the primary results and will remain accessible for 5 years.
Access Criteria: Access to de-identified IPD will be granted to qualified researchers with a methodologically sound proposal, subject to IRB approval and a signed data use agreement. Requests must be submitted via email to the principal investigator. Data will be shared through secure electronic means.
URL: https://www.imss.gob.mx/investigacion

REFERENCES:
- [Background] Basso A, Baldini P, Bertoldi G, Driussi G, Caputo I, Bettin E, Cacciapuoti M, Calo LA. Oxidative stress reduction by icodextrin-based glucose-free solutions in peritoneal dialysis: Support for new promising approaches. Artif Organs. 2024 Sep;48(9):1031-1037. doi: 10.1111/aor.14801. Epub 2024 Jun 1. PMID 38822597
- [Background] Kunin M, Beckerman P. The Peritoneal Membrane-A Potential Mediator of Fibrosis and Inflammation among Heart Failure Patients on Peritoneal Dialysis. Membranes (Basel). 2022 Mar 11;12(3):318. doi: 10.3390/membranes12030318. PMID 35323792
- [Background] Blake PG, Dong J, Davies SJ. Incremental peritoneal dialysis. Perit Dial Int. 2020 May;40(3):320-326. doi: 10.1177/0896860819895362. Epub 2020 Jan 17. PMID 32063212